CLINICAL TRIAL: NCT06767995
Title: Comparison of GlideScope® Titanium (Verathon) and Flexible Intubation Video Endoscope® (FIVE, Storz) In Terms Of Intubation Success In Infants With Pierre Robin Sequence
Brief Title: Comparison of Two Airway Devices in Paediatric Patients With Difficult Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Begum Ercan, Medical Doctor, Specialist, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HacettepeÜ-AR-BE-01
Record Dates: First submitted 2024-06-10; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Intubation; Difficult or Failed
Keywords: fiberoptic bronchoscope; videolaryngoscopy; difficult airway; Pierre Robin Sequence
MeSH Terms: conditions — Pierre Robin Syndrome

STUDY DESIGN:
Intervention Model Description: Our study is a prospective randomized controlled study. Intubation success and intubation times were compared with Flexible Intubation Video Endoscope (FIVE)® or GlideScope® Titanium devices in patients with Pierre Robin Sequence. Randomization was performed by a research assistant who used a computer to generate random numbers 1 and 2 and was terminated when the minimum number of patients in both groups was reached. The number 1 is assigned to the GlideScope® Titanium and the number 2 is assigned to the Flexible Intubation Video Endoscope® (FIVE). Randomization was concealed from the practitioner in a sealed envelope and informed to the practitioner after parental consent to participate in the study was obtained.
Who Masked: Care Provider
Masking Description: Patients were randomized and intubated by two experienced faculty members using either FFB or Glidescope. Intubation success on the first attempt, intubation duration, glottic visualization time, and complications were recorded by a non-blinded research assistant. Both devices were compared for these parameters.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intubation with Flexible fiberoptic bronchoscopy (Active Comparator): Patients were intubated with FFB and intubation success, intubation time, glottic visualization time and complications were recorded.
  FFB is considered the gold standard for airway management in both adult and pediatric patients with known or anticipated difficult airways.
  Interventions: Device: Flexible fiberoptic bronchoscopy
- Intubation with Glidescope (Active Comparator): Patients were intubated with Glidescope and intubation success, intubation time, glottic visualization time and complications were recorded.
  New generation videolaryngoscopy systems have also been successfully used as an alternative to FFB in pediatric patients with anticipated difficult airways. One of the most frequently used is Glidescope.
  Interventions: Device: Glidescope

INTERVENTIONS:
Device: Flexible fiberoptic bronchoscopy — If Flexible Intubation Video Endoscope® (FIVE) will be used, the appropriate endotracheal tube is loaded into the bronchoscope and made ready. The number of attempts and duration of successful intubation were recorded by a non-blinded research assistant. The stopwatch was started when the FFB started to pass through the patient's mouth/nose, and as soon as the ventilation of the lungs was confirmed by the end tidal carbon dioxide trace, the stopwatch was stopped and this time was recorded as the successful intubation time. The time between passing FFB through the mouth/nose and obtaining the best glottic view was recorded as the best glottic visualization time. The endotracheal tube passage time was defined as the intubation time minus the best glottic visualization time and recorded. Complications during the procedure were recorded.
  Other Names: Flexible Intubation Video Endoscope (FIVE)®
  Arms: Intubation with Flexible fiberoptic bronchoscopy
Device: Glidescope — If GlideScope® Titanium is to be used, a 50-60° angle is applied with the appropriate stylet, and the appropriate one from 3 pediatric blade sizes is selected according to the clinical experience of the relevant practitioner. The number of attempts and duration of successful intubation were recorded by a non-blinded research assistant. The stopwatch was started as soon as the videolaryngoscope started to pass through the patient's mouth, and the stopwatch was stopped as soon as the ventilation of the lungs was confirmed by the end tidal carbon dioxide trace, and this time was recorded as the successful intubation time. The time between passing the videolaryngoscope through the mouth/nose and obtaining the best glottic view was recorded as the best glottic visualization time. Endotracheal tube transit time was defined as intubation time minus best glottic visualization time and recorded. Complications during the procedure were recorded.
  Other Names: GlideScope® Titanium
  Arms: Intubation with Glidescope

SUMMARY:
The aim of current study was to compare Flexible fiberoptic bronchoscopy (FFB) and Glidescope devices in terms of intubation success and duration of intubation in patients under 12 months of age with PRS. In the present study, the investigators found similar initial intubation success rates with Glidescope and FFB. Although further studies are needed to determine the superiority of the two techniques, the investigators believes that advanced airway techniques should be prioritized and can be safely used by reducing the number of interventions.

DETAILED DESCRIPTION:
Flexible fiberoptic bronchoscopy (FFB) is considered the gold standard for airway management in both adult and pediatric patients with known or anticipated difficult airways. New generation videolaryngoscopy systems have also been successfully used as an alternative to FFB in pediatric patients with anticipated difficult airways. Airway management in patients with Pierre Robin Sequence (PRS) is challenging due to the classic triad of glossoptosis, micrognathia, and airway obstruction, along with potential accompanying syndromes and anomalies. It is clear that advanced airway techniques should be used in this patient group. However, there are not many studies in the literature demonstrating the success or superiority of these advanced airway techniques. The aim of current study was to compare FFB and Glidescope devices in terms of intubation success and duration of intubation in patients under 12 months of age with PRS. The current study is a prospective randomized controlled trial. Following ethical approval, between March 2021 and December 2023, intubation success and duration were compared between Flexible Intubation Video Endoscope (FIVE)® or GlideScope® Titanium devices in PRS patients under 12 months of age who underwent elective surgery under general anesthesia. Patients' anthropometric data such as age, weight, height, gender, preoperative airway examination measurements including mouth opening (MO), thyromental distance (TMD), frontal plane-chin distance (FPCD), and FPCD/weight index were recorded. Patients were randomized and intubated by two experienced faculty members using either FFB or Glidescope. Intubation success on the first attempt, intubation duration, glottic visualization time, and complications were recorded by a non-blinded research assistant. Both devices were compared for these parameters. The current study included 50 PRS patients, with 23 in the FFB group and 27 in the Glidescope group. There were no statistically significant differences between the two patient groups in terms of age, gender, anthropometric measurements, mouth opening, TMD, FPCD, and FPCD/weight index. There was no statistically significant difference in intubation success on the first attempt between the two groups (81.5% for Glidescope and 87% for FFB, p=0.430). The median intubation duration was statistically significantly shorter in the Glidescope group (35 seconds, IQR=10.5) compared to the FFB group (40 seconds, IQR=18) (p=0.032). Since the endotracheal tube passage times were similar in both groups, this difference was attributed to the time to achieve optimal glottic visualization. The median time to achieve optimal glottic visualization was 9.5 seconds (IQR=7.5) in the Glidescope group and 16 seconds (IQR=14) in the FFB group (p=0.002). However, the clinical significance of this difference cannot be conclusively determined. Moreover, complication rates during the procedure were similar between the two groups (18.5% for Glidescope and 13% for FFB, p=0.711). There is currently no validated test for predicting difficult preoperative airways in PRS patients. Literature reviews suggest that pediatric reference values for MO, TMD, and FPCD measurements are controversial, and more studies are needed to establish appropriate reference values. In the present study, the investigators found similar initial intubation success rates with Glidescope and FFB. Although further studies are needed to determine the superiority of the two techniques, the investigators believes that advanced airway techniques should be prioritized and can be safely used by reducing the number of interventions.

ELIGIBILITY:
Inclusion Criteria:

* Being under 12 months,
* Being diagnosed with Pierre Robin Sequence,
* Being subjected to elective surgery,
* To be operated between 01 March 2021 and 31 December 2023.

Exclusion Criteria:

* Patients requiring emergency surgery, patients requiring rapid serial intubation,
* Patients who have already been taken to the operating room by intubation or tracheostomy,
* Patients who will not be processed under general anesthesia,
* Patients who do not have family consent and informed consent cannot be obtained

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Intubation success on the first attempt | 34 months
  It was defined as a successful intubation attempt on the first attempt using FFB or Glidescope. Successful intubation was confirmed by end tidal carbon dioxide tracing. Failed intubation was defined as an intubation attempt lasting more than 120 seconds, removal and repositioning of the airway device from the mouth/nose, or esophageal intubation.

SECONDARY OUTCOMES:
Time to intubation | 34 months
  It is defined as the time between the FFB passing through the patient's mouth/nose or the videolaryngoscope passing through the patient's mouth and the end tidal carbon dioxide trace appearing on the monitor.
Glottic visualization time | 34 months
  It is defined as the time between the passage of the FFB through the patient's mouth/nose or the passage of the videolaryngoscope through the patient's mouth and the acquisition of the best glottic view.
Complications | 34 months
  Complications; esophageal intubation, desaturation defined as SpO2<90%, airway bleeding, soft tissue damage, bradycardia (heart rate below 90 beats/min), systolic hypotension (below 60mmHg for 0-1 months, below 70mmHg for 1-12 months), dysrhythmia was determined as cardiac arrest.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Medicine, Ankara, Sihhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT06767995/Prot_SAP_ICF_000.pdf